CLINICAL TRIAL: NCT01724931
Title: A Phase 2 Double-Blind, Placebo-Controlled, Randomized Dose Finding Study For The Efficacy And Safety Of Aminopterin In Methotrexate-Naive Rheumatoid Arthritis
Brief Title: Aminopterin Dose Finding Treatment for Methotrexate-Naïve Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Syntrix-AMT-RA-202
Record Dates: First submitted 2012-11-07; First posted 2012-11-12 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
Keywords: antifolate; antiinflammatory; autoimmune disease; hematological treatment; rheumatic disease; folic acid antagonist; enzyme inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo once weekly
  Interventions: Drug: placebo
- 3 mg LD-Aminopterin (Experimental): 3 mg LD-aminopterin once weekly
  Interventions: Drug: LD-aminopterin
- 1 mg LD-aminopterin (Experimental): 1 mg LD-aminopterin once weekly
  Interventions: Drug: LD-aminopterin

INTERVENTIONS:
Drug: LD-aminopterin
  Arms: 1 mg LD-aminopterin; 3 mg LD-Aminopterin
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether aminopterin is effective in the treatment of rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, dose ranging study that will evaluate the safety, efficacy, and pharmacokinetic properties (the absorption, distribution and excretion) of aminopterin following oral administration by subjects with active rheumatoid arthritis (≥ 6 tender and ≥ 6 swollen joints) who have not been treated with methotrexate (MTX). Subjects are randomized to one of three treatments: placebo, 1 mg of LD-aminopterin, or 3 mg of LD-aminopterin in a 1:1:1 ratio. The study hypothesis is that the 3 mg LD-aminopterin per week is effective at treating rheumatoid arthritis compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age.
2. A diagnosis of RA established by the ACR/EULAR 2010 criteria applied to patients who: 1) have >1 joint with definite clinical synovitis (swelling); 2) with the synovitis not better explained by another disease.

Add scores of categories A-D; a score >6/10 is required for study entry.

A. Joint involvement:

1 large joint=0; 2-10 large joints=1; 1-3 small joints (with or without involvement of large joints=2; 4-10 small joints (with or without involvement of large joints)=3; >10 joints (at least 1 small joint)=5.

B. Serology (at least 1 test result is needed for classification):

Negative RF and negative ACPA=0; Low-positive RF or low-positive ACPA=2; High-positive RF or high-positive ACPA=3.

C. Acute-phase reactants (at least 1 test result is needed for classification):

Normal CRP and normal ESR=0; Abnormal CRP or abnormal ESR=1.

D. Duration of symptoms:

less than 6 weeks=0; 6 weeks or greater=1.

3. Class I, II or III functional according to the ACR 1992 revised criteria for the classification of global functional status in RA.

4. RA is active, defined as ≥ 6 swollen joints and ≥ 6 tender joints.

5. Ability to understand and sign written informed consent.

6. For sexually active men and for women of childbearing potential, an adequate form of contraception.

7. For pre-menopausal women, a negative pregnancy test, obtained within 1 week prior to first study drug dose.

8. Negative serology for hepatitis B and hepatitis C.

9. The following screening laboratory blood tests must have the following values, or not clinically significant as determined by the PI and Medical Monitor: WBC WNL; absolute neutrophil count > lower limit of normal; platelet count WNL; hemoglobin >10.0 g/dL; AST WNL.

10. Adequate renal function: GFR estimated by Cockcroft-Gault formula >60 ml/min

Exclusion Criteria:

1. Known history of hepatitis, HIV infection, interstitial lung disease.
2. Alcohol consumption on a regular basis and unwilling, or unable, to discontinue this consumption during the study period.
3. Prior methotrexate or aminopterin therapy.
4. Prior biologic drug therapy (e.g., etanercept, adalimumab, infliximab).
5. Within 2 weeks prior to Study Day 0, or on Study Day 0, or at any time during the study, use of any of the following medications that may result in drug/drug interactions with AMT: trimethoprim with or without sulfamethoxazole; sulfonamides; sulfonylureas; pyrimethamine; triamethamine; dipyridamole; colchicine; probenecid; aminoglycosides; theophylline; phenytoin; and folinic acid (i.e., leucovorin).
6. At Study Day 0 use of DMARDs and biologics (except antimalarials) including oral or injectable gold, azathioprine, penicillamine, sulfasalazine or cyclosporine. Subjects previously treated with any of these medications are eligible provided a 28 day wash-out is completed prior to Study Day 0. Antimalarial can be continued at the same dose if they have been administered at the same dose for 8 weeks before Study Day 0, and they will be administered at the same dose throughout the study. NSAIDs or corticosteroid (≤ 10 mg prednisone or equivalent/day) may be continued at the same dose if they have been used at a stable dose for two weeks prior to Study Day 0, and will be continued at the same doses throughout the study.
7. Use of corticosteroids in excess of 10 mg prednisone or equivalent/day.
8. Known concurrent malignancy except basal or squamous cell skin carcinoma, or cervical carcinoma in situ.
9. Concurrent participation in another clinical trial involving experimental treatment within 30 days of Study Day 0.
10. Current and uncontrolled infection, cardiovascular, renal, pulmonary, hepatic or GI conditions that will interfere with the conduct of the trial or pose a morbid risk.
11. Investigator's opinion that a concurrent disease or condition impairs the subject's ability to complete the trial: includes psychological, familial, sociological, geographical or medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
ACR20 | Study Day 84
  The primary efficacy endpoint, determined at study day 84 or last observation carried forward (LOCF), is the percent of subjects who obtain ACR20 in the 3 mg/week LD-AMT dose compared to placebo.

SECONDARY OUTCOMES:
ACR20 | Study Day 84
  A secondary efficacy endpoint, determined at study day 84 or LOCF, is the percent of subjects who obtain ACR20 in the 1 mg LD-AMT/week dose.

OTHER OUTCOMES:
Adverse Event | Study Day 126
  Adverse events, including laboratory measurements of serum chemistry and hematology, and the occurrence of dose-limiting toxicity. Safety endpoints will be evaluated throughout the study and for an additional 42 days after a subject goes off study.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Kahn, MD, MS, Study Director — Syntrix Biosystems, Inc.
Locations (15):
- Ukraine (15):
  - Centre of Immunobiologic Therapy, State Institution "Institute of Emergency and Reconstructive Surgery, Donets'k
  - Department of Hospital Therapy #1, Regional Clinical Hospital for occupational diseases 104, Donetsk
  - Communal Establishment of Health Protection, Regional Hospital of Veterans of War, Rheumatology Department, Kharkiv
  - Department of Rheumatology, Communal Establishment of Health Protection "Kharkiv City Clinical Hospital #8", Kharkiv
  - National Scientific Center "M.D. STRAZHESKO INSTITUTE OF CARDIOLOGY, MAS OF UKRAINE", Kyiv
  - Department of Rheumatology and Allergology, Kyiv Regional Clinical Hospital №1, Kyiv
  - Lviv Regional Clinical Hospital, Department of Rheumatology, Lviv
  - Department of Cardio-Rheumatology, Communal Institution "Odesa Regional Clinical Hospital", Odesa
  - Crimean State Medical University n.a. S.I. Georgievsky based on Rheumatology Department of Crimean Republic Institution "Clinical Territorial Medical Association "University Clinic", Simferopol
  - Railway Clinical Hospital of Uzhorod Station of Lviv Railroad Administration, Therapeutic Department, Uzhhorod
  - Department of Rheumatology, Vinnytsya Regional Clinical Hospital n.a. M.I, Vinnytsa
  - Zaporizhzhya City Multiple Discipline Clinical Hospital #9, Department of Therapy, Zaporizhzhya
  - Department of Rheumatology, Zaporizhzhia Regional Clinical Hospital, Zaporizhzhya
  - Department of Therapy, City Clinical Hospital № 6, Zaporizhzhya
  - Department of Therapy, City Hospital № 7, Zaporizhzhya

REFERENCES:
- [Result] Menter A, Thrash B, Cherian C, Matherly LH, Wang L, Gangjee A, Morgan JR, Maeda DY, Schuler AD, Kahn SJ, Zebala JA. Intestinal transport of aminopterin enantiomers in dogs and humans with psoriasis is stereoselective: evidence for a mechanism involving the proton-coupled folate transporter. J Pharmacol Exp Ther. 2012 Sep;342(3):696-708. doi: 10.1124/jpet.112.195479. Epub 2012 May 31. PMID 22653877